CLINICAL TRIAL: NCT02304523
Title: A Prospective, Randomized, Single-blinded (Evaluator), 3-treatment Arm, Parallel, Multi-center, Phase 3 Trial to Evaluate Safety and Efficacy of CDFR0612 and CDFR0613
Brief Title: Safety and Efficacy of CDFR0612 and CDFR0613 for Bowel Cleansing Before Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CTC Bio, Inc. (Industry)
Collaborators: Symyoo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTC-BCS-CDFR0612/0613_3
Record Dates: First submitted 2014-11-27; First posted 2014-12-02 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Colonoscopy Preparation; Colon Disease
Keywords: Colonoscopy preparation; Bowel cleansing; Colon cleansing; Colonoscopy; CDFR0612; CDFR0613
MeSH Terms: conditions — Colonic Diseases | interventions — MoviPrep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test 1 (Experimental): CDFR0612 Solution 150mL will be mixed with water of 350ml to prepare a bowel cleansing preparation solution 500mL. Take it within 30min. After then, take additional water 500ml within 30min.
  These processes will be in evening at one day before colonoscopy and in early morning at the same day of colonoscopy.
  Interventions: Drug: CDFR0612
- Test 2 (Experimental): CDFR0613 Solution 150mL will be mixed with water of 350ml to prepare a bowel cleansing preparation solution 500mL. Take it within 30min. After then, take additional water 500ml within 30min.
  These processes will be in evening at one day before colonoscopy and in early morning at the same day of colonoscopy.
  Interventions: Drug: CDFR0613
- Comparator (Active Comparator): Coolprep Powder A and B will be mixed with water to prepare a mixture of a bowel cleansing preparation solution 500mL. Repeat it twice. Take these of IL (2 * 500mL) within 1 hour. After then, take additional 500ml water.
  These processes will be in evening at one day before colonoscopy and in early morning at the same day of colonoscopy.
  Interventions: Drug: Coolprep Powder

INTERVENTIONS:
Drug: CDFR0612 — Preparation 500mL is a mixture of CDFR0612 150mL and water 350mL. A total of 2L (Preparation 1L and additional water 1L) will be administrated divided into two in evening before and in early morning at that day of colonoscopy.
  Arms: Test 1
Drug: CDFR0613 — Preparation 500mL is a mixture of CDFR0613 150mL and water 350mL. A total of 2L (Preparation 1L and additional water 1L) will be administrated divided into two in evening before and in early morning at that day of colonoscopy.
  Arms: Test 2
Drug: Coolprep Powder — Preparation 500mL is a water solution of Coolprep Powder A and B. A total of 3L (Preparation 2L and additional water 1L) will be administrated divided into two in evening before and in early morning at that day of colonoscopy.
  Other Names: Moviprep
  Arms: Comparator

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of CDFR0612 and CDFR0613 compared to PEG+picosulfate (Coolprep Powder) preparation. The effectiveness for bowel cleansing will be assessed with Harefield Cleansing Scale (HCS) by blinded assessor.

DETAILED DESCRIPTION:
This study is a prospective, randomized, single-blinded, parallel, 3-treatment, multi-center clinical trial. A total of 297 subjects scheduled for colonoscopy will participate to this study and be assigned to 3 groups - CDFR0612, CDFR0613, or a comparator (Coolprep Powder). A subject will admit to hospital one day before colonoscopy and be administrated with study drug. In early morning at the that day of colonoscopy, he/she will be administrated with study drug again. Any subject will be carefully monitored for safety during hospitalisation (1 night) and additional 4 weeks follow-up period because this study is the first human trial of CDFR0612 and CDFR0613.

ELIGIBILITY:
Inclusion Criteria:

* Patients who is informed and give a consent in voluntary
* Patients who is scheduled a colonoscopy
* BMI 19≤ and <30

Exclusion Criteria:

* Patients who participate in other interventional study or had participated within 30 days before screening
* Pregnant or breast-feeding women who do not want to stop breast-feeding
* Women of childbearing potential who do not agree with appropriate contraception during this study
* Patients who had experienced any hypersensitivity study drug or ingredient
* Uncontrolled hypertension
* Arrhythmia with clinically significant findings from EKG
* Congestive heart failure; NYHA functional class III or IV; unstable coronary artery disease; myocardiac infarction history within 6 months
* Uncontrolled diabetes
* Active infection except acute upper respiratory infection or local skin infection; Fever (38 °C and higher) within 1 week before study administration
* HIV infection and/or chronic hepatitis B or C
* Patients who has a difficulty to participate because of severe nausea or vomiting
* Suspected or confirmed inflammatory bowel disease, toxic colon or toxic megacolon, or gastrointestinal obstruction or perforation; visible bleeding in colon
* History of colon surgery and abdominal surgery within 6 month; need an emergency surgery
* Colonoscopy for the following use: treatment of bleeding from such lesions as vascular malformation, ulceration, neoplasia, and polypectomy site (e.g.,electrocoagulation, heater probe, laser or injection therapy); foreign body removal; decompression of acute nontoxic megacolon or sigmoid volvulus; balloon dilation of stenotic lesions (e.g., anastomotic strictures); palliative treatment of stenosing or bleeding neoplasms (e.g., laser, electrocoagulation, stenting)
* Fluid or electrolyte (Na, K, Ca, Mg, chloride, bicarbonate) disturbance
* Severe dehydration risk (e.g., rhabdomyolysis, ascites)
* Dialysis or renal disorder (creatinine clearance <15ml/min)
* Suspected pulmonary aspiration or gag reflex disorder
* History of hypersensitivity of drug or others
* Alcohol or drug abuse within 6 months
* Clinically significant underlying disease or medical history at investigator's discretion
* Inability in written/verbal communication

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Successful cleansing rate | post-colonoscopy at Day 2
  %Patient with HCS-graded A or B

SECONDARY OUTCOMES:
Overall cleansing rate | post-colonoscopy at Day 2
  %Patient with each HCS-grade (A, B, C, D)
Mean segmental cleansing score | post-colonoscopy at Day 2
  5 Segment: Rectum, Sigmoid colon, Descending colon, Transverse colon, Ascending colon/cecum.
Patient reported outcomes | Post-dosing at Day 1 and Day 2
  Patient questionnaire about any patient discomfort related to study drug administration
Cecal intubation rate | post-colonoscopy at Day 2
Mean cecal intubation time | post-colonoscopy at Day 2
Mean colonoscopy withdrawal time | post-colonoscopy at Day 2
Treatment Compliance | Post dosing at Day 2
Polyp detection rate | post-colonoscopy at Day 2

OTHER OUTCOMES:
Treatment-emergent adverse events | For 4 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Woo KIM, M.D., Principal Investigator — Seoul St. Mary's Hospital; Dongjin Yoo, M.D., Study Director — Symyoo
Locations (4):
- South Korea (4):
  - Uijengbu St.Mary's Hospital, Uijengbu-si, Gyeonggi-do
  - Seoul St.Mary's Hospital, Seoul, Seocho-gu, Banpo-daero
  - Korea University Anam Hospital, Seongbuk-gu, Seoul
  - Korea University Ansan Hospital, Ansan